CLINICAL TRIAL: NCT00135226
Title: A Study of Cardiovascular Events iN Diabetes - A Randomized 2x2 Factorial Study of Aspirin Versus Placebo, and of Omega-3 Fatty Acid Supplementation Versus Placebo, for Primary Prevention of Cardiovascular Events in People With Diabetes
Brief Title: ASCEND: A Study of Cardiovascular Events iN Diabetes
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other); Bayer (Industry); Medical Research Council (Other Government); Solvay Pharmaceuticals (Industry); Abbott (Industry); Mylan (Unknown); Health Data Research UK (Unknown); Alzheimer's Research UK (Unknown); The Macular Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTSUASCEND1; 60635500 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Cardiovascular Disease; Aspirin; Omega-3 fatty acids; Primary prevention; Randomized Controlled Trial; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; n-3 fatty acid
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Aspirin; Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Aspirin + Omega-3 Ethyl Esters (Active Comparator): Participants receive 100mg of aspirin once daily and 1g of omega-3 ethyl esters once daily.
  Interventions: Drug: Aspirin; Drug: Omega-3 Ethyl Esters
- Aspirin + Placebo Omega-3 Ethyl Esters (Active Comparator): Participants receive 100mg of aspirin once daily and placebo omega-3 ethyl esters once daily.
  Interventions: Drug: Aspirin; Drug: Placebo Omega-3 Ethyl Esters
- Placebo Aspirin + Omega-3 Ethyl Esters (Active Comparator): Participants receive placebo aspirin once daily and 1g of omega-3 ethyl esters once daily.
  Interventions: Drug: Omega-3 Ethyl Esters; Drug: Placebo Aspirin
- Placebo Aspirin + Placebo Omega-3 Ethyl Esters (Active Comparator): Participants receive placebo aspirin once daily and placebo omega-3 ethyl esters once daily.
  Interventions: Drug: Placebo Aspirin; Drug: Placebo Omega-3 Ethyl Esters

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin + Omega-3 Ethyl Esters; Aspirin + Placebo Omega-3 Ethyl Esters
Drug: Omega-3 Ethyl Esters
  Other Names: n-3 fatty acid; Omacor
  Arms: Aspirin + Omega-3 Ethyl Esters; Placebo Aspirin + Omega-3 Ethyl Esters
Drug: Placebo Aspirin
  Arms: Placebo Aspirin + Omega-3 Ethyl Esters; Placebo Aspirin + Placebo Omega-3 Ethyl Esters
Drug: Placebo Omega-3 Ethyl Esters
  Arms: Aspirin + Placebo Omega-3 Ethyl Esters; Placebo Aspirin + Placebo Omega-3 Ethyl Esters

SUMMARY:
The purpose of this study is to determine whether 100mg daily aspirin versus placebo and/or supplementation with 1 gram daily omega-3 fatty acids or placebo prevents "serious vascular events" (i.e. non-fatal heart attack, non-fatal stroke or transient ischaemic attack, or death from vascular causes) in patients with diabetes who are not known to have occlusive arterial disease and to assess the effects on serious bleeding or other adverse events.

DETAILED DESCRIPTION:
The role of antiplatelet therapy (chiefly aspirin) for the secondary prevention of heart attacks and strokes is firmly established for many high-risk people with diagnosed arterial disease, and the proportional reductions in these cardiovascular events appear to be about one quarter, whether or not such patients have diabetes. But, most younger and middle-aged people with diabetes do not have manifest arterial disease - although they are still at significant cardiovascular risk - and yet few trials have tested aspirin in such individuals. As a result, there is substantial uncertainty about the role of aspirin for the prevention of heart attacks and strokes among apparently healthy people with diabetes, and only a small minority receives it.

There is consistent evidence from observational studies of lower rates of cardiovascular disease (particularly cardiac and sudden death) in people with higher intakes, or higher blood levels, of fish oils (omega-3 fatty acids). Trials in people who have survived a heart attack have shown modest, but potentially worthwhile, reductions in coronary events.

If ASCEND can reliably demonstrate that aspirin and/or fish oils safely reduce the risk of cardiovascular events and deaths in people with diabetes who do not have pre-existing arterial disease, then this would be relevant to some tens of millions of people world-wide (who are currently not receiving such therapy) and might save tens of thousands of lives each year.

The initial results (published 2018) showed that aspirin prevented serious vascular events in patients with diabetes who did not already have cardiovascular disease, but it caused almost as many major bleeds and there was no effect on cancers. There was no significant difference in the risk of serious vascular events between those who were assigned to receive n-3 fatty acid supplementation and those who were assigned to receive placebo.

ASCEND will be conducting long-term follow-up for 20-years beyond the scheduled treatment period (which ended in 2017). We will collect relevant data from UK central health registries. This will be used to assess whether the balance of benefits versus hazards of aspirin observed within the main trial, relating to major vascular events such as heart attack or stroke, continue long-term or whether additional benefits emerge during longer-term follow-up.

In addition ASCEND will use this long-term post-trial follow-up to investigate further whether low-dose aspirin might protect against cancer. The main cancer analyses is planned to take place ~5-years after the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with type 1 or type 2 diabetes mellitus.
* Aged ≥ 40 years.
* No previous history of vascular disease.
* No clear contra-indication to aspirin.
* No other predominant life-threatening medical problem.

Exclusion Criteria:

* Definite history of myocardial infarction, stroke or arterial revascularisation procedure.
* Currently prescribed aspirin, warfarin or any other blood thinning medication.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15480 (Actual)
Dates: Start 2005-03; Primary Completion 2018-03-12 (Actual); Study Completion 2037-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jane M Armitage, BSc, MBBS, MRCP, FFPH, Principal Investigator — Clinical Trial Service Unit, NDPH, University of Oxford
Locations (1):
- Clinical Trial Service Unit, NDPH, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Proposals for substudies must be approved by the Steering Committee. Procedures for accessing the data for this study are available on: https://www.ndph.ox.ac.uk/about/data-access-policy.
Supporting Information: Study Protocol, SAP
Access Criteria: See URL
URL: https://www.ndph.ox.ac.uk/about/data-access-policy

REFERENCES:
- [Background] Harper C, Mafham M, Herrington W, Staplin N, Stevens W, Wallendszus K, Haynes R, Landray MJ, Parish S, Bowman L, Armitage J. Comparison of the Accuracy and Completeness of Records of Serious Vascular Events in Routinely Collected Data vs Clinical Trial-Adjudicated Direct Follow-up Data in the UK: Secondary Analysis of the ASCEND Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2139748. doi: 10.1001/jamanetworkopen.2021.39748. PMID 34962561
- [Background] Harper C, Mafham M, Herrington W, Staplin N, Stevens W, Wallendszus K, Haynes R, Landray MJ, Parish S, Bowman L, Armitage J. Reliability of major bleeding events in UK routine data versus clinical trial adjudicated follow-up data. Heart. 2023 Sep 13;109(19):1467-1472. doi: 10.1136/heartjnl-2023-322616. PMID 37270201
- [Background] Sammons E, Bowman L, Stevens W, Buck G, Wallendszus K, Hammami I, Parish S, Armitage J; ASCEND Collaborative Group. ASCEND-Eye: Rationale, design and baseline characteristics for a sub-study of the ASCEND randomised trial, exploring the effects of aspirin and omega-3 fatty acids on diabetic retinopathy and age-related macular degeneration. Contemp Clin Trials Commun. 2023 Jul 5;35:101184. doi: 10.1016/j.conctc.2023.101184. eCollection 2023 Oct. PMID 37745288
- [Result] Parish S, Mafham M, Offer A, Barton J, Wallendszus K, Stevens W, Buck G, Haynes R, Collins R, Bowman L, Armitage J. Effects of aspirin on dementia and cognitive function in diabetic patients: the ASCEND trial. Eur Heart J. 2022 Jun 1;43(21):2010-2019. doi: 10.1093/eurheartj/ehac179. PMID 35393614
- [Result] Parish S, Mafham M, Offer A, Barton J, Wallendszus K, Stevens W, Buck G, Haynes R, Collins R, Bowman L, Armitage J; ASCEND Study Collaborative Group. Effects of Omega-3 Fatty Acid Supplements on Arrhythmias. Circulation. 2020 Jan 28;141(4):331-333. doi: 10.1161/CIRCULATIONAHA.119.044165. Epub 2020 Jan 27. No abstract available. PMID 31986094
- [Result] ASCEND Study Collaborative Group; Bowman L, Mafham M, Wallendszus K, Stevens W, Buck G, Barton J, Murphy K, Aung T, Haynes R, Cox J, Murawska A, Young A, Lay M, Chen F, Sammons E, Waters E, Adler A, Bodansky J, Farmer A, McPherson R, Neil A, Simpson D, Peto R, Baigent C, Collins R, Parish S, Armitage J. Effects of Aspirin for Primary Prevention in Persons with Diabetes Mellitus. N Engl J Med. 2018 Oct 18;379(16):1529-1539. doi: 10.1056/NEJMoa1804988. Epub 2018 Aug 26. PMID 30146931
- [Result] ASCEND Study Collaborative Group; Bowman L, Mafham M, Wallendszus K, Stevens W, Buck G, Barton J, Murphy K, Aung T, Haynes R, Cox J, Murawska A, Young A, Lay M, Chen F, Sammons E, Waters E, Adler A, Bodansky J, Farmer A, McPherson R, Neil A, Simpson D, Peto R, Baigent C, Collins R, Parish S, Armitage J. Effects of n-3 Fatty Acid Supplements in Diabetes Mellitus. N Engl J Med. 2018 Oct 18;379(16):1540-1550. doi: 10.1056/NEJMoa1804989. Epub 2018 Aug 26. PMID 30146932
- [Result] Bowman L, Mafham M, Stevens W, Haynes R, Aung T, Chen F, Buck G, Collins R, Armitage J; ASCEND Study Collaborative Group. ASCEND: A Study of Cardiovascular Events iN Diabetes: Characteristics of a randomized trial of aspirin and of omega-3 fatty acid supplementation in 15,480 people with diabetes. Am Heart J. 2018 Apr;198:135-144. doi: 10.1016/j.ahj.2017.12.006. Epub 2017 Dec 24. PMID 29653635
- [Result] Sammons EL, Buck G, Bowman LJ, Stevens WM, Hammami I, Parish S, Armitage J; ASCEND Study Collaborative Group. ASCEND-Eye: Effects of Omega-3 Fatty Acids on Diabetic Retinopathy. Ophthalmology. 2024 May;131(5):526-533. doi: 10.1016/j.ophtha.2023.11.030. Epub 2023 Dec 3. PMID 38052385
- [Result] Sammons EL, Buck G, Bowman LJ, Stevens WM, Hammami I, Parish S, Armitage J; ASCEND Study Collaborative Group. ASCEND-Eye: Effects of Aspirin on Diabetic Retinopathy. Ophthalmology. 2024 Jul;131(7):771-779. doi: 10.1016/j.ophtha.2024.01.018. Epub 2024 Jan 17. PMID 38237868
- [Result] Petrucci G, Buck GA, Rocca B, Parish S, Baigent C, Hatem D, Mafham M, Habib A, Bowman L, Armitage J, Patrono C. Thromboxane biosynthesis and future events in diabetes: the ASCEND trial. Eur Heart J. 2024 Apr 14;45(15):1355-1367. doi: 10.1093/eurheartj/ehad868. PMID 38385506
- [Result] Sammons E, Bowman L, Stevens W, Buck G, Hammami I, Parish S, Armitage J; ASCEND-Eye Collaborative Group. Effects of aspirin and omega-3 fatty acids on age-related macular degeneration in ASCEND-Eye: a randomised placebo-controlled trial in a population with diabetes. BMJ Open. 2025 Feb 26;15(2):e090605. doi: 10.1136/bmjopen-2024-090605. PMID 40010818
- [Result] Sammons EL, Buck G, Bowman LJ, Stevens WM, Hammami I, Parish S, Armitage J; ASCEND Study Collaborative Group. Effects of aspirin and omega-3 fatty acids on composite and subdomain scores from the NEI-VFQ-25 questionnaire: the ASCEND-Eye randomized controlled trial. BMC Ophthalmol. 2024 Nov 5;24(1):481. doi: 10.1186/s12886-024-03741-x. PMID 39501183
- [Derived] Parish S, Buck G, Aung T, Mafham M, Clark S, Hill MR, Collins R, Bowman L, Armitage J; ASCEND Study Collaborative Group. Effect of low-dose aspirin on urinary 11-dehydro-thromboxane B2 in the ASCEND (A Study of Cardiovascular Events iN Diabetes) randomized controlled trial. Trials. 2023 Mar 4;24(1):166. doi: 10.1186/s13063-023-07198-z. PMID 36871000
- See also: The study website for information about ASCEND: A Study of Cardiovascular Events iN Diabetes — https://www.ctsu.ox.ac.uk/research/ascend

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized between June 2005 through July 2011. Follow-up continued until March 2018.
Groups:
- Aspirin + Omega-3 Ethyl Esters: Participants receive 100mg of aspirin once daily and 1g of omega-3 ethyl esters once daily.
  Aspirin
  Omega-3 ethyl esters
- Aspirin + Placebo Omega-3 Ethyl Esters: Participants receive 100mg of aspirin once daily and placebo omega-3 ethyl esters once daily.
  Aspirin
  Placebo omega-3 ethyl esters
- Placebo Aspirin + Omega-3 Ethyl Esters: Participants receive placebo aspirin once daily and 1g of omega-3 ethyl esters once daily.
  Placebo aspirin
  Omega-3 ethyl esters
- Placebo Aspirin + Placebo Omega-3 Ethyl Esters: Participants receive placebo aspirin once daily and placebo omega-3 ethyl esters once daily.
  Placebo aspirin
  Placebo omega-3 ethyl esters
Period: Overall Study
Arm/Group | Aspirin + Omega-3 Ethyl Esters | Aspirin + Placebo Omega-3 Ethyl Esters | Placebo Aspirin + Omega-3 Ethyl Esters | Placebo Aspirin + Placebo Omega-3 Ethyl Esters
Started | 3870 | 3870 | 3870 | 3870
Completed | 3836 | 3835 | 3836 | 3834
Not Completed | 34 | 35 | 34 | 36

BASELINE CHARACTERISTICS:
Groups:
- Aspirin + Omega-3: Participants receive 100mg of aspirin once daily and 1g of omega-3 ethyl esters once daily.
- Aspirin + Placebo Omega-3: Participants receive 100mg of aspirin once daily and placebo omega-3 ethyl esters once daily.
- Placebo Aspirin + Omega-3: Participants receive placebo aspirin once daily and 1g of omega-3 ethyl esters once daily.
- Placebo Aspirin + Placebo Omega-3: Participants receive placebo aspirin once daily and placebo omega-3 ethyl esters once daily.
- Total: Total of all reporting groups
Arm/Group | Aspirin + Omega-3 | Aspirin + Placebo Omega-3 | Placebo Aspirin + Omega-3 | Placebo Aspirin + Placebo Omega-3 | Total
Number analyzed (Participants) | 3870 | 3870 | 3870 | 3870 | 15480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2257 | 2259 | 2257 | 2261 | 9034
  >=65 years | 1613 | 1611 | 1613 | 1609 | 6446
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.3) | 63.2 (9.1) | 63.3 (9.2) | 63.3 (9.2) | 63.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1448 | 1449 | 1450 | 1449 | 5796
  Male | 2422 | 2421 | 2420 | 2421 | 9684
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic origin: White | 3733 | 3734 | 3734 | 3734 | 14935
  Ethnic origin: Indian/Pakistani/Bangladeshi | 46 | 45 | 46 | 47 | 184
  Ethnic origin: African/Caribbean | 34 | 36 | 36 | 34 | 140
  Ethnic origin: Other/unknown | 57 | 55 | 54 | 55 | 221
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3870 | 3870 | 3870 | 3870 | 15480
Body-mass index (kg/m²) [Count of Participants; unit: Participants] — The body-mass index (the weight in kilograms divided by the square of the height in meters) was based on values for weight and height that were reported by the participants.
  Participants
    <25 | 522 | 558 | 607 | 562 | 2249
    ≥25 to <30 | 1356 | 1397 | 1415 | 1361 | 5529
    ≥30 | 1863 | 1802 | 1721 | 1815 | 7201
    Unknown | 129 | 113 | 127 | 132 | 501
Body-mass index (mean) [Mean (Standard Deviation); unit: kg/m²] | 30.9 (6.3) | 30.8 (6.2) | 30.5 (6.3) | 30.7 (6.3) | 30.7 (6.3)
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 319 | 320 | 320 | 320 | 1279
  Ex-smoker | 1764 | 1762 | 1763 | 1762 | 7051
  Never smoked | 1745 | 1744 | 1744 | 1744 | 6977
  Unknown | 42 | 44 | 43 | 44 | 173
Treated hypertension [Count of Participants; unit: Participants] — Participant reported hypertension
  Participants
    Yes | 2384 | 2382 | 2384 | 2383 | 9533
    No | 1459 | 1460 | 1458 | 1458 | 5835
    Unknown | 27 | 28 | 28 | 29 | 112
Aspirin use prior to screening [Count of Participants; unit: Participants]
  Yes | 1373 | 1367 | 1371 | 1397 | 5508
  No | 2497 | 2503 | 2499 | 2473 | 9972
Type of diabetes [Count of Participants; unit: Participants] — The presence of type 2 diabetes was based on a broad clinical definition involving the age of the participant at the diagnosis of diabetes, the use of insulin within 1-year after diagnosis, and the body-mass index.
  Participants
    Type 1 | 226 | 232 | 234 | 219 | 911
    Type 2 | 3644 | 3638 | 3636 | 3651 | 14569
Duration of diabetes (years) [Count of Participants; unit: Participants]
  <6 yr | 2172 | 2165 | 2160 | 2162 | 8659
  ≥6 <13 yr | 1484 | 1492 | 1496 | 1493 | 5965
  ≥13 yr | 214 | 213 | 214 | 215 | 856
Duration of diabetes (years) [Median (Inter-Quartile Range); unit: years] | 7 [3 to 13] | 7 [3 to 13] | 7 [3 to 12] | 7 [3 to 13] | 7 [3 to 13]
Systolic blood pressure (mmHg) [Count of Participants; unit: Participants]
  <130 mmHg | 849 | 845 | 846 | 854 | 3394
  ≥130 to <140 mmHg | 764 | 786 | 783 | 758 | 3091
  ≥140 mmHg | 1140 | 1123 | 1139 | 1153 | 4555
  Unknown | 1117 | 1116 | 1102 | 1105 | 4440
Systolic blood pressure (mean) [Mean (Standard Deviation); unit: mmHg] | 136.1 (15.4) | 136.1 (15.0) | 136.2 (15.3) | 136.2 (15.2) | 136.2 (15.3)
Vascular risk score [Count of Participants; unit: Participants] — We categorized the predicted 5-year risk of serious vascular event (including transient ischemic attack) without the use of aspirin or n-3 fatty acids as follows: low risk as less than 5%, moderate risk as 5% to less than 10%, and high risk as 10% or more.
  Participants
    Low (<5%) | 1567 | 1561 | 1577 | 1559 | 6264
    Moderate (≥5%, <10%) | 1635 | 1659 | 1634 | 1620 | 6548
    High (≥10%) | 668 | 650 | 659 | 691 | 2668

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Any Serious Vascular Event (SVE)
Description: The primary efficacy assessments involve intention-to-treat comparisons among all randomized participants of allocation to aspirin versus placebo and, separately, of omega-3 fatty acids versus placebo on the first occurrence of any "Serious Vascular Event" (SVE), defined as:
  * non-fatal myocardial infarction; or
  * non-fatal stroke (excluding confirmed intracranial hemorrhage) or TIA; or
  * vascular death excluding confirmed intracranial hemorrhage (defined as International Classification of Diseases 10th revision [ICD-10] I00-52 or I63-99, i.e. excluding subarachnoid hemorrhage [I60], intracerebral hemorrhage [I61], and other non-traumatic intracranial hemorrhage [I62]).
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Groups:
- Aspirin: Group includes 3870 participants in the Aspirin+Omega-3 arm, and 3870 participants in the Aspirin+Placebo Omega-3 arm
- Placebo Aspirin: Group includes 3870 participants in the Placebo Aspirin+Omega-3 arm, and 3870 participants in the Placebo Aspirin+Placebo Omega-3 arm
- Omega-3: Group includes 3870 participants in the Omega-3+Aspirin arm, and 3870 participants in the Omega-3+Placebo Aspirin arm
- Placebo Omega-3: Group includes 3870 participants in the Placebo Omega-3+Aspirin arm, and 3870 participants in the Placebo Omega-3+Placebo Aspirin arm
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 658 | 743 | 689 | 712
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; p = 0.01, Log Rank; Rate Ratio = 0.88, 95% CI 2-sided [0.79 to 0.97]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; p = 0.55, Log Rank; Rate Ratio = 0.97, 95% CI 2-sided [0.87 to 1.08]

2. Primary Outcome: Number of Participants With First Occurrence of Any Major Bleed (Aspirin Comparison Only)
Description: The primary safety assessments involve intention-to-treat comparisons among all randomized patients of allocation to aspirin versus placebo on the first occurrence of "any major bleed", defined as:
  * any confirmed intracranial hemorrhage (including intracerebral, subarachnoid, subdural or any other intracranial hemorrhage); or
  * sight-threatening eye bleeding; or
  * any other serious bleeding episode.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin
Number analyzed (Participants) | 7740 | 7740
Participants | 314 | 245
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; p = 0.003, Log Rank; Rate Ratio = 1.29, 95% CI 2-sided [1.09 to 1.52]

3. Secondary Outcome: Number of Participants With Combined End-point of Serious Vascular Events (SVEs) or Revascularizations
Description: Secondary efficacy assessments involve intention-to-treat comparisons among all randomized participants of allocation to aspirin versus placebo and, separately, of omega-3 versus placebo on the first occurrence of the expanded vascular endpoint of "SVE or revascularization" (including coronary and non-coronary revascularizations).
Time Frame: Randomized treatment phase during a mean of 7.4 years
Population: A single participant may have had multiple events.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 833 | 936 | 882 | 887
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.88, 95% CI 2-sided [0.80 to 0.97]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 1.00, 95% CI 2-sided [0.91 to 1.09]

4. Secondary Outcome: Number of Participants With Any Incident Gastrointestinal (GI) Tract Cancer (Aspirin Comparison Only)
Description: Secondary efficacy assessments of aspirin involve intention-to-treat comparisons during the scheduled treatment period among all randomized participants on the first occurrence of:
  Any incident gastrointestinal (GI) tract cancer (i.e. any GI cancer excluding pancreas and hepatobiliary), overall and after exclusion of the first three years of follow-up.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Population: Participants taking aspirin
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin
Number analyzed (Participants) | 7740 | 7740
Participants | 157 | 158
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.99, 95% CI 2-sided [0.80 to 1.24]

5. Other Pre Specified Outcome: Number of Participants With Fatal Event: All-cause Mortality
Description: 'All-cause mortality' includes all recorded deaths.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 748 | 792 | 752 | 788
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.94, 95% CI 2-sided [0.85 to 1.04]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Risk Ratio = 0.95, 95% CI 2-sided [0.86 to 1.05]

6. Other Pre Specified Outcome: Number of Participants With Fatal Event: Coronary
Description: Fatal 'Coronary' events include deaths from: Acute MI and other CHD (unspecified Acute ischaemic heart disease; Atherosclerotic heart disease; Ischaemic cardiomyopathy; unspecified Chronic ischaemic heart disease).
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 105 | 122 | 100 | 127
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.86, 95% CI 2-sided [0.66 to 1.12]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate ratio = 0.79, 95% CI 2-sided [0.61 to 1.02]

7. Other Pre Specified Outcome: Number of Participants With Fatal Event: All Stroke
Description: Fatal 'All stroke' events include deaths from: Haemorrhagic stroke (Intracerebral haemorrhage; Subarachnoid haemorrhage); Non-haemorrhagic stroke (Cerebral infarction; Stroke not specified as haemorrhage or infarction).
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 38 | 34 | 35 | 37
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 1.12, 95% CI 2-sided [0.7 to 1.77]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 0.94, 95% CI 2-sided [0.59 to 1.50]

8. Other Pre Specified Outcome: Number of Participants With Fatal Event: Other Vascular
Description: Fatal 'Other vascular' events include deaths from: Heart failure (excluding ischaemic cardiomyopathy); Other vascular death (excluding stroke; and Cardiac death (excluding CHD).
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 67 | 70 | 61 | 76
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.96, 95% CI 2-sided [0.68 to 1.34]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 0.80, 95% CI 2-sided [0.57 to 1.12]

9. Other Pre Specified Outcome: Number of Participants With Fatal Event: Cancer
Description: Fatal 'Cancer' events include any death attributed to cancer.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 309 | 315 | 305 | 319
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.98, 95% CI 2-sided [0.84 to 1.15]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate ratio = 0.95, 95% CI 2-sided [0.82 to 1.12]

10. Other Pre Specified Outcome: Number of Participants With Fatal Event: Respiratory
Description: Fatal 'Respiratory' events include any death attributed to respiratory causes.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 82 | 69 | 73 | 78
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate ratio = 1.19, 95% CI 2-sided [0.86 to 1.63]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 0.93, 95% CI 2-sided [0.68 to 1.28]

11. Other Pre Specified Outcome: Number of Participants With Fatal Event: Other Medical
Description: Fatal 'Other medical' events include deaths from: Non-vascular medical causes (excluding cancer and respiratory, including Fatal GI bleed or perforation); and deaths from Renal disease and Diabetes.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 126 | 157 | 158 | 125
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.80, 95% CI 2-sided [0.64 to 1.01]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 1.26, 95% CI 2-sided [1.00 to 1.59]

12. Other Pre Specified Outcome: Number of Participants With Fatal Event: External Cause
Description: Fatal 'External cause' events include deaths from: Injury; Fracture; Self harm; and Medical and surgical complications
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 18 | 21 | 17 | 22
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.86, 95% CI 2-sided [0.46 to 1.60]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate ratio = 0.77, 95% CI 2-sided [0.41 to 1.45]

13. Other Pre Specified Outcome: Number of Participants With Fatal Event: Unknown Cause
Description: Any death for which the cause is not known.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 3 | 4 | 3 | 4
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.75, 95% CI 2-sided [0.17 to 3.30]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 0.75, 95% CI 2-sided [0.17 to 3.31]

14. Other Pre Specified Outcome: Number of Participants With Event: Any Cancer
Description: Incidence of fatal or non-fatal cancers. Any cancer excludes non-fatal non-melanoma skin cancer and non-fatal recurrence of a cancer that had occurred before randomization.
  A single participant may have had multiple cancers.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 897 | 887 | 894 | 890
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 1.01, 95% CI 2-sided [0.92 to 1.11]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Risk Ratio = 1.00, 95% CI 2-sided [0.91 to 1.10]

15. Other Pre Specified Outcome: Number of Participants With Event: Other Gastrointestinal Cancer (Aspirin Comparison Only)
Description: Includes fatal and non-fatal cancers. Excludes cancers reported in the gastrointestinal tract category (see secondary outcome measure #4), and includes hepatobiliary and pancreatic cancers.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin
Number analyzed (Participants) | 7740 | 7740
Participants | 87 | 82
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 1.06, 95% CI 2-sided [0.78 to 1.43]

16. Other Pre Specified Outcome: Number of Participants With Event: Respiratory Cancer
Description: Includes fatal and non-fatal cancers. Includes lung and larynx cancer.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 101 | 103 | 104 | 100
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate ratio = 0.98, 95% CI 2-sided [0.74 to 1.29]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 1.04, 95% CI 2-sided [0.79 to 1.37]

17. Other Pre Specified Outcome: Number of Participants With Event: Genitourinary Cancer
Description: Includes fatal and non-fatal renal, bladder, prostate, gynaecological and other GU cancers
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 332 | 294 | 323 | 303
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 1.13, 95% CI 2-sided [0.97 to 1.32]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 1.07, 95% CI 2-sided [0.91 to 1.25]

18. Other Pre Specified Outcome: Number of Participants With Event: Hematological Cancer
Description: Includes fatal and non-fatal cancers. Includes leukaemia and lymphoma.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 88 | 86 | 94 | 80
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 1.02, 95% CI 2-sided [0.76 to 1.38]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 1.17, 95% CI 2-sided [0.87 to 1.58]

19. Other Pre Specified Outcome: Number of Participants With Event: Breast Cancer
Description: Includes fatal and non-fatal cancers.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 97 | 96 | 103 | 90
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 1.01, 95% CI 2-sided [0.76 to 1.34]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 1.14, 95% CI 2-sided [0.86 to 1.52]

20. Other Pre Specified Outcome: Number of Participants With Event: Melanoma
Description: Includes fatal and non-fatal melanomas.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 50 | 59 | 55 | 54
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.85, 95% CI 2-sided [0.58 to 1.23]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate ratio = 1.02, 95% CI 2-sided [0.70 to 1.48]

21. Other Pre Specified Outcome: Number of Participants With Event: Other Cancer
Description: Includes fatal and non-fatal cancers not included elsewhere (where the type of cancer is known).
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 25 | 30 | 23 | 32
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.83, 95% CI 2-sided [0.49 to 1.41]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 0.72, 95% CI 2-sided [0.42 to 1.22]

22. Other Pre Specified Outcome: Number of Participants With Event: Unspecified Cancer
Description: Includes fatal and non-fatal cancers of unknown type.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740 | 7740 | 7740
Participants | 26 | 31 | 25 | 32
Statistical Analysis 1: Comparison: Aspirin vs Placebo Aspirin; Test type: Other; Rate Ratio = 0.84, 95% CI 2-sided [0.50 to 1.41]
Statistical Analysis 2: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 0.78, 95% CI 2-sided [0.46 to 1.31]

23. Other Pre Specified Outcome: Number of Participants With Event: Atrial Fibrillation (Omega-3 Comparison Only)
Description: Includes fatal and non-fatal events.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740
Participants | 166 | 135
Statistical Analysis 1: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 1.23, 95% CI 2-sided [0.98 to 1.54]

24. Other Pre Specified Outcome: Number of Participants With Event: Other Arrhythmia (Omega-3 Comparison Only)
Description: Includes fatal and non-fatal events, excludes atrial fibrillation.
Time Frame: Randomized treatment phase during a mean of 7.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 | Placebo Omega-3
Number analyzed (Participants) | 7740 | 7740
Participants | 83 | 99
Statistical Analysis 1: Comparison: Omega-3 vs Placebo Omega-3; Test type: Other; Rate Ratio = 0.84, 95% CI 2-sided [0.63 to 1.12]

ADVERSE EVENTS:
Time Frame: Randomized treatment phase during a mean of 7.4 years
Description: Follow-up questionnaires asking about cardiovascular events and other Serious Adverse Events were sent to participants at 6-monthly intervals.
  Only information about Serious Adverse Events were collected, therefore there are no Non-Serious Adverse Events to report.
Arm/Group | Aspirin | Placebo Aspirin | Omega-3 | Placebo Omega-3
All-Cause Mortality (participants affected / at risk) | 748/7740 | 792/7740 | 752/7740 | 788/7740
Serious Adverse Events (participants affected / at risk) | 5264/7740 | 5321/7740 | 5344/7740 | 5241/7740
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin (N=7740) | Placebo Aspirin (N=7740) | Omega-3 (N=7740) | Placebo Omega-3 (N=7740)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 184 | 145 | 156 | 173
Cardiac disorders (Cardiac disorders) | 784 | 824 | 812 | 796
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 5 | 4 | 6 | 3
Ear and labyrinth disorders (Ear and labyrinth disorders) | 44 | 15 | 23 | 36
Endocrine disorders (Endocrine disorders) | 21 | 21 | 24 | 18
Eye disorders (Eye disorders) | 511 | 457 | 486 | 482
Gastrointestinal disorders (Gastrointestinal disorders) | 664 | 635 | 671 | 628
General disorders and administration site conditions (General disorders) | 240 | 231 | 247 | 224
Hepatobiliary disorders (Hepatobiliary disorders) | 112 | 149 | 134 | 127
Immune system disorders (Immune system disorders) | 27 | 19 | 16 | 30
Infections and infestations (Infections and infestations) | 859 | 804 | 847 | 816
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 484 | 479 | 488 | 475
Investigations (Investigations) | 906 | 965 | 935 | 936
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 200 | 176 | 201 | 175
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 248 | 256 | 265 | 239
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1320 | 1266 | 1294 | 1292
Nervous system disorders (Nervous system disorders) | 724 | 776 | 741 | 759
Psychiatric disorders (Psychiatric disorders) | 35 | 41 | 36 | 40
Renal and urinary disorders (Renal and urinary disorders) | 381 | 384 | 387 | 378
Reproductive system and breast disorders (Reproductive system and breast disorders) | 157 | 130 | 137 | 150
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 436 | 351 | 395 | 392
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 171 | 127 | 131 | 167
Social circumstances (Social circumstances) | 2 | 2 | 3 | 1
Surgical and medical procedures (Surgical and medical procedures) | 2916 | 2990 | 2990 | 2916
Vascular disorders (Vascular disorders) | 192 | 213 | 194 | 211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT00135226/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT00135226/SAP_000.pdf